CLINICAL TRIAL: NCT04211415
Title: DS-2741a Phase I Study- A Three-part First-in-human Study: Single Ascending Dose and Multiple Dose Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of DS-2741a After Subcutaneous Injection in Healthy Japanese Male Subjects, and Single Dose Study to Assess the Pharmacokinetics, Safety, Pharmacodynamics and Efficacy of DS-2741a After Subcutaneous Injection in Japanese Subjects With Moderate to Severe Atopic Dermatitis.
Brief Title: Phase I Study of DS-2741a in Healthy Volunteers and Participants With Atopic Dermatitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision of termination of the clinical program.
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DS2741-A-J101; 195071 (Other: JapicCTI ID)
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; DS-2741a
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant, care provider, investigator, and outcomes assessor will be blinded in Part 1 and Part 3 of the study. Part 2 of the study will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Part 1: DS-2741a Cohort 1, 5 mg (Experimental): Participants will be randomized to receive a single, subcutaneous injection of DS-2741a 5 mg.
  Interventions: Drug: DS-2741a
- Part 1: DS-2741a Cohort 2, 15 mg (Experimental): Participants will be randomized to receive a single, subcutaneous injection of DS-2741a 15 mg.
  Interventions: Drug: DS-2741a
- Part 1: DS-2741a Cohort 3, 50 mg (Experimental): Participants will be randomized to receive a single, subcutaneous injection of DS-2741a 50 mg.
  Interventions: Drug: DS-2741a
- Part 1: DS-2741a Cohort 4, 150 mg (Experimental): Participants will be randomized to receive a single, subcutaneous injection of DS-2741a 150 mg.
  Interventions: Drug: DS-2741a
- Part 1: DS-2741a Cohort 5, 500 mg (Experimental): Participants will be randomized to receive a single, subcutaneous injection of DS-2741a 500 mg.
  Interventions: Drug: DS-2741a
- Part 1: DS-2741a Cohort 6, 1000 mg (Experimental): Participants will be randomized to receive a single, subcutaneous injection of DS-2741a 1000 mg.
  Interventions: Drug: DS-2741a
- Part 1: Placebo (Placebo Comparator): Participants will be randomized to receive a single, subcutaneous injection of placebo.
  Interventions: Drug: Placebo
- Part 2: DS-2741a Cohort 1, X mg (based on results of Part 1) (Experimental): Participants will receive a single, subcutaneous injection of DS-2741a X mg, where X mg will be based on the maximum tolerated dose identified in Part 1.
  Interventions: Drug: DS-2741a
- Part 2: DS-2741a Cohort 1, Y mg (based on results of Part 1) (Experimental): Participants will receive a single, subcutaneous injection of DS-2741a Y mg, where Y mg will be based on the maximum tolerated dose identified in Part 1.
  Interventions: Drug: DS-2741a
- Part 3: DS-2741a Cohort 1, Z mg (based on results of Part 1) (Experimental): Participants will be randomized to receive a receive a single, subcutaneous injection of DS-2741a Z mg, where Z mg will be based on the maximum tolerated dose identified in Part 1.
  Interventions: Drug: DS-2741a
- Part 3: Placebo (Placebo Comparator): Participants will be randomized to receive a single, subcutaneous injection of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DS-2741a — Single, subcutaneous injection (upper arm, upper part of the thigh, or abdominal wall in principle) administered weekly for 4 weeks
  Arms: Part 1: DS-2741a Cohort 1, 5 mg; Part 1: DS-2741a Cohort 2, 15 mg; Part 1: DS-2741a Cohort 3, 50 mg; Part 1: DS-2741a Cohort 4, 150 mg; Part 1: DS-2741a Cohort 5, 500 mg; Part 1: DS-2741a Cohort 6, 1000 mg; Part 2: DS-2741a Cohort 1, X mg (based on results of Part 1); Part 2: DS-2741a Cohort 1, Y mg (based on results of Part 1); Part 3: DS-2741a Cohort 1, Z mg (based on results of Part 1)
Drug: Placebo — Single, subcutaneous injection administered weekly for 4 weeks
  Arms: Part 1: Placebo; Part 3: Placebo

SUMMARY:
This is a phase 1, single-center, first-in-human study to assess the safety, pharmacokinetics and pharmacodynamics of DS-2741a after subcutaneous injection in healthy Japanese male volunteers and Japanese participants with moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
This study consists of three parts. Part 1 and Part 3 are a single ascending and multiple dose study to assess the safety, pharmacokinetics and pharmacodynamics of DS-2741a after subcutaneous injection in healthy Japanese male participants. Part 2 is a single-dose study to assess the pharmacokinetics, safety, pharmacodynamics and efficacy of DS-2741a after subcutaneous injection in Japanese participants with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* For Part 1 and Part 3:

  * Japanese healthy male subjects.
  * Age ≥20 and ≤45 years upon providing informed consent.
  * Body mass index (BMI) ≥18.5 and <25.0 kg/m^2 at screening.
* For Part 2:

  * Japanese Male or female, Age ≥20 upon providing informed consent.
  * Diagnosed with chronic atopic dermatitis (AD) at least 3 years before screening and by the criteria of Hannifin and Rajka at screening.

Exclusion Criteria:

* For Part 1 and Part 3:

  * Having a history of atopic dermatitis
  * Having a history of hypersensitivity to drugs or other substances or being idiosyncratic
  * Having alcohol or drug dependence, etc.
* For Part 2:

  * Having an active dermatological disease other than AD, which, in the investigator's opinion, would affect study assessments.
  * Having a history of serious disease in the study potentially endangering the participant, as judged by the investigator or sub-investigator.
  * Having a chronic or acute infection requiring treatment within 28 days before screening.
  * Having superficial skin infections within 7 days before screening.
  * Having a history of recurrent oral herpes and recurrent genital herpes.
  * Having a history of parasitic infection or invasive, opportunistic infection such as histoplasmosis despite infection resolution, etc.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events among participants receiving DS-2741a (Part 1 and Part 3) | Day 1 through end of study, up to 4 weeks
Characterize pharmacokinetic parameter maximum plasma concentration (Cmax) of plasma DS-2741a (Part 2) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 11, Day 14, Day 17, Day 21, Day 28, Day 35, Day 42, Day 49
Characterize pharmacokinetic parameter time to reach maximum plasma concentration (Tmax) of plasma DS-2741a (Part 2) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 11, Day 14, Day 17, Day 21, Day 28, Day 35, Day 42, Day 49
Characterize pharmacokinetic parameter area under the curve from time 0 to last measurable time point (AUClast) of plasma DS-2741a (Part 2) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 11, Day 14, Day 17, Day 21, Day 28, Day 35, Day 42, Day 49
Characterize pharmacokinetic parameter area under the curve from time 0 to 168 h (AUC168h) of plasma DS-2741a (Part 2) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 11, Day 14, Day 17, Day 21, Day 28, Day 35, Day 42, Day 49
Characterize pharmacokinetic parameter total clearance (CL/F) of plasma DS-2741a (Part 2) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 11, Day 14, Day 17, Day 21, Day 28, Day 35, Day 42, Day 49
Characterize pharmacokinetic parameter area under the curve from time 0 to infinity (AUCinf) of plasma DS-2741a (Part 2) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 11, Day 14, Day 17, Day 21, Day 28, Day 35, Day 42, Day 49
Characterize pharmacokinetic parameter terminal elimination half-life (t1/2) of plasma DS-2741a (Part 2) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 11, Day 14, Day 17, Day 21, Day 28, Day 35, Day 42, Day 49
Characterize pharmacokinetic parameter volume of distribution (Vz/F) of plasma DS-2741a (Part 2) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 11, Day 14, Day 17, Day 21, Day 28, Day 35, Day 42, Day 49

SECONDARY OUTCOMES:
Characterize pharmacokinetic parameter maximum plasma concentration (Cmax) of plasma DS-2741a (Part 1) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 11, Day 14, Day 17, Day 21, Day 28, Day 35, Day 42, Day 49
Characterize pharmacokinetic parameter time to reach maximum plasma concentration (Tmax) of plasma DS-2741a (Part 1) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 11, Day 14, Day 17, Day 21, Day 28, Day 35, Day 42, Day 49
Characterize pharmacokinetic parameter area under the curve from time 0 to last measurable time point (AUClast) of plasma DS-2741a (Part 1) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 11, Day 14, Day 17, Day 21, Day 28, Day 35, Day 42, Day 49
Characterize pharmacokinetic parameter area under the curve from time 0 to 168 h (AUC168h) of plasma DS-2741a (Part 1) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 11, Day 14, Day 17, Day 21, Day 28, Day 35, Day 42, Day 49
Characterize pharmacokinetic parameter total clearance (CL/F) of plasma DS-2741a (Part 1) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 11, Day 14, Day 17, Day 21, Day 28, Day 35, Day 42, Day 49
Characterize pharmacokinetic parameter area under the curve from time 0 to infinity (AUCinf) of plasma DS-2741a (Part 1) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 2, Day 3, Day 4,Day 5, Day 6, Day 7, Day 8, Day 9, Day 11, Day 14, Day 17, Day 21, Day 28, Day 35, Day 42, Day 49
Characterize pharmacokinetic parameter terminal elimination half-life (t1/2) of plasma DS-2741a (Part 1) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 11, Day 14, Day 17, Day 21, Day 28, Day 35, Day 42, Day 49
Characterize pharmacokinetic parameter volume of distribution (Vz/F) of plasma DS-2741a (Part 1) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 11, Day 14, Day 17, Day 21, Day 28, Day 35, Day 42, Day 49
Incidence of anti-drug antibodies (ADAs) against DS-2741a (Part 1 and Part 2) | Day 1 (pre-dose), Day 28, Day 49
Incidence of adverse events among participants receiving DS-2741a (Part 2) | Day 1 through end of study, up to 4 weeks
Characterize pharmacokinetic parameter maximum plasma concentration (Cmax) of plasma DS-2741a (Part 3) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 3, Day 5, Day 7 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 10, Day 12, Day 14 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 17
Characterize pharmacokinetic parameter time to reach maximum plasma concentration (Tmax) of plasma DS-2741a (Part 3) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 3, Day 5, Day 7 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 10, Day 12, Day 14 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 17
Characterize pharmacokinetic parameter trough plasma concentration (Ctrough) of plasma DS-2741a (Part 3) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 3, Day 5, Day 7 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 10, Day 12, Day 14 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 17
Characterize pharmacokinetic parameter area under the curve from time 0 to 168 h (AUC168h) of plasma DS-2741a (Part 3) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 3, Day 5, Day 7 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 10, Day 12, Day 14 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 17
Characterize pharmacokinetic parameter area under the curve from time 0 to tau (504-672 h) (AUCtau) of plasma DS-2741a (Part 3) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 3, Day 5, Day 7 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 10, Day 12, Day 14 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 17
Characterize pharmacokinetic parameter terminal elimination half-life (t1/2) of plasma DS-2741a (Part 3) | Day 1 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 3, Day 5, Day 7 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 10, Day 12, Day 14 (pre-dose, 2, 8, 24, 36 hours after the start of administration), Day 17
Incidence of anti-drug antibodies (ADAs) against DS-2741a (Part 3) | Day 1 (pre-dose),Day 7 (pre-dose), Day 14 (pre-dose), Day 21 (pre-dose), Day 49, Day 63

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (1):
- Osaka Pharmacology Clinical Research Hospital, Osaka, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://www.vivli.org/ourmember/daiichi-sankyo/